CLINICAL TRIAL: NCT01108328
Title: A Prospective, Single Crossover, Randomized, Double Blind Placebo Controlled Trial Evaluating Subjective Ratings of Appetite and Glucoregulation of a Low Calorie Diet Supplemented With a High Viscosity Polysaccharide (PolyGlycopleX - PGX) vs. Rice Flour Control, in Overweight and Moderately Obese Females.
Brief Title: Evaluation of Subjective Ratings of Appetite and Glucoregulation of a Low Calorie Diet Supplemented With a High Viscosity Polysaccharide (PolyGlycopleX - PGX)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Center for Functional Medicine (Other)
Collaborators: University of British Columbia (Other); InovoBiologic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PGX Crossover Study
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Appetite and Hunger, Suppression; Blood Glucose, Postprandial
Keywords: viscous; fibre; polysaccharide; blood glucose; postprandial; appetite; hunger; satiety
MeSH Terms: interventions — PolyGlycoplex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- PolyGlycopleX (PGX) (Experimental): 5 grams of PGX 3 times per day with each main meal (breakfast, lunch and dinner)
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)
- Rice flour (Placebo Comparator): 5 grams of rice flour 3 times per day at each main meal (breakfast, lunch and dinner)
  Interventions: Dietary Supplement: PolyGlycopleX (PGX)

INTERVENTIONS:
Dietary Supplement: PolyGlycopleX (PGX) — powder, 5 grams, 3 times per day at each main meal (breakfast, lunch and dinner) for a total of 3 days

SUMMARY:
The objective of the study is to compare subjective appetite ratings and after-meal and 24 hour blood glucose levels within overweight and obese female subjects consuming either a standardized 3 day low calorie diet supplemented with a viscous fibre known as PGX (treatment) or a rice flour (placebo control). Each treatment phase will be 3 days in length and separated by 3 week washout phase, so subjects will also be acting as their own control. Subjects will be randomized to either start with the low calorie diet with PGX or the low calorie diet supplemented with rice flour. We hypothesize that the 3 day LCD with PGX will elicit an improved appetite score compared to the 3 day LCD supplemented with the rice flour placebo control.

ELIGIBILITY:
Inclusion Criteria:

- BMI 25-35 Kg/m2

Exclusion Criteria:

* Known diabetes
* Medications or natural health products that affect appetite
* Contraindications to LCD
* Any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the protocol.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in the ratings of the variables in the Appetite Visual Analog Scale and the overall Appetite Score. | 3 days

SECONDARY OUTCOMES:
Changes in 2-hour postprandial areas under the curve (AUC) and 24 hour blood glucose (CGMS) profiles. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lyon, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Canadian Centre for Functional Medicine, Coquitlam, British Columbia
  - Canadian Center for Functional Medicine, Coquitlam, British Columbia

REFERENCES:
- [Result] Kacinik V, Lyon M, Purnama M, Reimer RA, Gahler R, Green TJ, Wood S. Effect of PGX, a novel functional fibre supplement, on subjective ratings of appetite in overweight and obese women consuming a 3-day structured, low-calorie diet. Nutr Diabetes. 2011 Dec 12;1(12):e22. doi: 10.1038/nutd.2011.18. PMID 23154443